CLINICAL TRIAL: NCT05203926
Title: Significance and Outcome of Magnetic Resonance Enterography Revealing Sacroiliitis in Crohn's Disease: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Spondyloarthritis Research and Treatment Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-00955
Record Dates: First submitted 2021-12-23; First posted 2022-01-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Sacroiliitis
MeSH Terms: conditions — Sacroiliitis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crohn's disease (CD) subjects (Experimental): These subjects will then undergo T1 and STIR sequence MRI of SI joints (pelvis MRI) as well as SIJ plain X-ray for assessment of radiographic sacroiliitis.
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — Subjects will undergo T1 and STIR sequence MRI of sacroiliac joints (SIJ ) (pelvis MRI) as well as SIJ plain X-ray for assessment of radiographic sacroiliitis. The study will utilize 3 Tesla with phased array coil to maximize signal to noise ratio for image quality. This is a single procedure, which takes about 60 minutes. 1 radiologists, blinded to all clinical information, will evaluate for presence of acute and structural lesions. Images will be scored for presence or absence of acute and/or structural lesions in a global manner.

SUMMARY:
This study aims to further define and characterize imaging findings of possible sacroiliitis in Crohn's Disease patients by recalling subjects who had findings of possible sacroiliitis on prior MRE and assess the natural history and outcome of these cases by using standard magnetic resonance imaging (MRI) and x-ray of the sacroiliac joints.

DETAILED DESCRIPTION:
When axial spondyloarthritis (SpA) occurs in Crohn's disease (CD) is an important clinical and research question that has not been fully answered. Magnetic resonance enterography (MRE), routinely obtained in Crohn's disease (CD) patients, can be utilized to assess sacroiliac joints (SIJ); currently published literature shows that it could be a valuable tool to detect active inflammation of sacroiliitis in CD patients. Only a small fraction of CD patients with MRE evidence of sacroiliitis is referred to rheumatologists for further evaluation. The proposed project aims to further define MRE features of sacroiliitis in CD by recalling subjects who had prior positive findings and assess the natural history and outcome of these cases by standard magnetic resonance imaging (MRI) of sacroiliac joints and SIJ X-ray. 37 CD subjects who were already found to have sacroiliitis in the previous MRE study will be recalled. Subjects will undergo standard MRI of SIJ, plain X-ray of SIJ and the rheumatologist will obtain detailed history and examine patients for evaluation of possible axial SpA. Other details pertaining to CD, CD therapy and activity, will also be obtained to help clarify a correlation between CD and axial SpA. This pilot study will allow better characterization of imaging features of sacroiliitis on MRE, provide useful information on clinical significance of these lesions in CD patients, and potentially establish MRE as a screening tool for early detection of sacroiliitis in CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of sacroiliitis on earlier standard of care MRE between 2014 and 2018.
* Confirmed diagnosis of Crohn's Disease
* Known HLA-B27 status at time of enrollment and most recent clinical ESR and CRP results from chart (from day of visit or within past 4 weeks of study visit)
* Adults >18 years of age

Exclusion Criteria:

* History of other inflammatory arthritis (e.g. rheumatoid arthritis, systemic lupus erythematosus, gout).
* Contraindication to MRI.
* History of malignancy <5 years in remission, (except for non-melanomatous skin cancer).
* Inability to comply with study protocol.
* Critically ill patients.
* Pregnant patients.
* Non-English speaking patients (as the questionnaires used in this study are not validated in other languages)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Significance of sacroiliitis features/lesions seen on Magnetic Resonance Enterography (MRE) | Intervention Visit 1 (Day 1)
  The MRI scans will establish significance of sacroiliitis features/lesions seen on MRE.
Significance of sacroiliitis features/lesions seen on Magnetic Resonance Enterography (MRE) | Intervention Visit 1 (Day 1)
  The X-ray exams will establish significance of sacroiliitis features/lesions seen on MRE.

SECONDARY OUTCOMES:
Measurement of Ankylosing Spondylitis Disease Activity | Intervention Visit 1 (Day 1)
  ASDAS- Ankylosing Spondylitis Disease Activity Score will assesses patient-perceived symptoms and current disease activity through serum markers. The higher the score the higher the disease activity.
Measurement of Bath Ankylosing Spondylitis Disease Activity Index | Intervention Visit 1 (Day 1)
  BASDAI- Bath Ankylosing Spondylitis Disease Activity Index assesses Ankylosing Spondylitis Disease activity and current symptoms. The BASDAI sum score is calculated by the sum of questions 1-4 plus mean of questions 5 and 6, the total then divided by 5. The sum score ranges from 0 to 10, higher values indicate more active disease.
Measurement of Bath Ankylosing Spondylitis Functional Index | Intervention Visit 1 (Day 1)
  BASFI- Bath Ankylosing Spondylitis Functional Index assesses functional limitation in patients with Ankylosing Spondylitis. The patient rates his/her ability to perform tasks (BASFI) by marking a vertical line on a 100 mm horizontal line. It consists of ten tasks lines to assess the degree of difficulty of performing each task. The total BASFI score is calculated by adding all ten scores and dividing by 10.
Measurement of HBI- Harvey-Bradshaw Index | Intervention Visit 1 (Day 1)
  HBI- Harvey-Bradshaw Index measures clinical activity of Crohn's Disease. The categorical HBI score was also used as an independent variable in all analyses. Specifically, HBI < 5 was defined as clinical remission, HBI between 5 and 7 as mild disease, HBI between 8 and 16 as moderate disease, and HBI > 16 as severe disease.
Measurement of CDAI- Crohn's Disease Activity Index | Intervention Visit 1 (Day 1)
  CDAI- Crohn's Disease Activity Index determines current severity of Crohn's Disease. CDAI scores range from 0 to 600. A score of less than 150 corresponds to relative disease quiescence (remission); 150 to 219, mildly active disease; 220 to 450, moderately active disease; and greater than 450, severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Fardina Malik, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data collected from this study include anthropomorphic and blood draw data that will be uploaded to the participants' EHR and questionnaire data that will only be used for study-related purposes